CLINICAL TRIAL: NCT03902288
Title: Fresh Pomegranate Juice Decreases Fasting Serum Erythropoietin in Patients With Type 2 Diabetes
Brief Title: Short-term Effect of Pomegranate Juice on Blood Sugar and Its Controlling Hormones in Pre-diabetic and Type II Diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Saleem A. Banihani, Associate Professor Doctor, Jordan University of Science and Technology
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20120189
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Patients With Type 2 Diabetes (FSG: More Than 7.1 and Not Higher Than 15.8 mmol/L)
Keywords: Patients with type 2 diabetes; Fresh pomegranate juice; Fasting serum glucose

STUDY DESIGN:
Intervention Model Description: A Patient with type 2 diabetes ( < 15.8 FSG) and healthy individual ingested fresh pomegranate at 1.5 mL per kg of body weight after approximately 12 hours fasting. Blood samples were collected before (- 5 min) and after 1 and 3 hours of ingesting pomegranate juice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with type 2 diabetes (Experimental): Patients with type 2 diabetes at early stages of type 2 diabetes (FSG: 7.1 15.8 mmol/L)
  Interventions: Other: Fresh pomegranate juice
- Healthy individuals (Active Comparator): Healthy individuals match age and gender to the experimental group
  Interventions: Other: Fresh pomegranate juice

INTERVENTIONS:
Other: Fresh pomegranate juice — Pomegranate seeds (arils) were separated by hand, and fresh pomegranate juice was prepared by squeezing the seeds using a fruit squeezing machine. Fresh pomegranate juice was given at 1.5 mL/kg of body weight for the fasted recruited patient with type 2 diabetes (FSG < 15.8 mmol/L). Blood was collected before and after 1 and 3 hours of ingesting the juice.

SUMMARY:
Fresh pomegranate juice at 1.5 mL/kg of body weight was administered by recruited healthy individuals and patients with type 2 diabetes of fasting serum glucose between 7.1 and 15.8 mmol/L after approximately 12 hours fasting. Blood samples were collected in plain tubes before (-5 minutes) and at 1 and 3 hours after drinking pomegranate juice. Blood samples were centrifuged and serum was collected and stored for glucose and hormonal analysis. Patients were recruited from those of earlier stages of type 2 diabetes, and many of them already drink pomegranate juice as of its benefits for their health).

The exclusion criteria included subjects with renal or hepatic disease, pregnancy, treatment with insulin, and hormone therapies. Participants who had either smoked cigarettes or taken antioxidant supplements, lipid-lowering drugs, and oral hypoglycemic agents, such as metformin (glucophage) or sulfonylureas, within the preceding 12 hours were also excluded.

The study was explained to all of the recruited subjects by the clinical researchers, and written informed consent was obtained prior to enrollment. Approval for the study was provided by the IRB Committee at Jordan University of Science and Technology (Irbid, Jordan).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes at early stages of progression (Fasting serum glucose: 7.1 - 15.8 mmol/L)
* Healthy individuals (Fasting serum glucose < 7 mmol/L)

Exclusion Criteria:

* Subjects with renal
* Subjects with hepatic disease
* Pregnant women
* Subjects under treatment with insulin and any other hormonal therapies
* Smoking 12 hours before the intervention
* Antioxidant supplements 12 hours before the intervention
* Drugs administration: Lipid lowering drugs, oral hypoglycemic agents such as metformin or sulfonylureas 12 hours before the intervention.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Fasting serum glucose measurement | 1 - 3 hours
  Measuring the alteration in fasting serum glucose in mmol/L before and at 1 and 3 hours following pomegranate juice ingestion
Insulin hormone measurement | 1 - 3 hours
  Measuring insulin in μIU/mL before and at 1 and 3 hours following pomegranate juice ingestion
Erythropoietin hormone measurement | 1 - 3 hours
  Measuring erythropoietin in mIU/mL before and at 1 and 3 hours following pomegranate juice ingestion
Thyroxine hormone measurement | 1 - 3 hours
  Measuring erythropoietin in μg/dL before and at 1 and 3 hours following pomegranate juice ingestion
Cortisol hormone measurement | 1 -3 hours
  Measuring erythropoietin in nmol/L before and at 1 and 3 hours following pomegranate juice ingestion

SECONDARY OUTCOMES:
Melatonin hormone measurement | 1 - 3 hours
  Measuring Melatonin in pg/mL before and at 1 and 3 hours following pomegranate juice ingestion
Testosterone hormone measurement | 1 - 3 hours
  Measuring testosterone in ng/dL before and at 1 and 3 hours following pomegranate juice ingestion
Aldosterone hormone measurement | 1 - 3 hours
  Measuring aldosterone in ng/dL before and at 1 and 3 hours following pomegranate juice ingestion
Serum total antioxidant activity measurement | 1 - 3 hours
  Measuring serum total antioxidant activity in Trolox equivalents before and at 1 and 3 hours following pomegranate juice ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Saleem A. Banihani, PHD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banihani SA, Shuaibu SM, Al-Husein BA, Makahleh SS. Fresh Pomegranate Juice Decreases Fasting Serum Erythropoietin in Patients with Type 2 Diabetes. Int J Food Sci. 2019 Apr 18;2019:1269341. doi: 10.1155/2019/1269341. eCollection 2019. PMID 31139640